CLINICAL TRIAL: NCT04700072
Title: A Phase 1/2 Open-Label Rolling-Arm Umbrella Platform Design of Investigational Agents With or Without Pembrolizumab or Pembrolizumab Alone in Participants With Melanoma (KEYMAKER-U02): Substudy 02D
Brief Title: Substudy 02D: Safety and Efficacy of Pembrolizumab in Combination With Investigational Agents or Pembrolizumab Alone in Participants With Melanoma Brain Metastasis (MK-3475-02D/KEYMAKER-U02)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-02D; MK-3475-02D (Other: MSD); KEYMAKER-U02 (Other: MSD); 2023-506315-17-00 (Registry Identifier: EU CT); U1111-1293-5704 (Registry Identifier: UTN); 2020-003742-36 (EudraCT Number)
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Melanoma
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Coformulation Pembrolizumab/Quavonlimab + Lenvatinib (Experimental): Participants will receive pembrolizumab/quavonlimab (coformulation of pembrolizumab and quavonlimab) intravenously (IV) plus lenvatinib orally at specified doses on specified days for a total treatment duration of up to approximately 2 years.
  Interventions: Biological: Pembrolizumab; Biological: Pembrolizumab/Quavonlimab; Drug: Lenvatinib
- Pembrolizumab + Lenvatinib (Experimental): Participants will receive pembrolizumab IV plus lenvatinib orally at specified doses on specified days for a total treatment duration of up to approximately 2 years.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — Administered via IV infusion at a specified dose on specified days
  Other Names: MK-3475; KEYTRUDA®
Biological: Pembrolizumab/Quavonlimab — Administered via IV infusion at a specified dose on specified days
  Other Names: MK-1308A
  Arms: Coformulation Pembrolizumab/Quavonlimab + Lenvatinib
Drug: Lenvatinib — Administered via oral capsule at a specified dose on specified days
  Other Names: MK-7902; E7080; LENVIMA®

SUMMARY:
Substudy 02D is part of a larger research study that is testing experimental treatments for melanoma, a type of skin cancer. The larger study is the umbrella study.

The goal of substudy 02D is to evaluate the safety and efficacy of investigational treatment arms in programmed cell-death 1 (PD-1) naïve or PD-1 exposed participants with melanoma brain metastasis (MBM) and to identify the investigational agent(s) that, when used in combination, are superior to the current treatment options/historical control available.

As of amendment 2 (effective 01DEC2022) enrollment into the treatment arm of pembrolizumab and lenvatinib has been discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Has American Joint Committee on Cancer (AJCC) Stage IV, M1D melanoma
* Is neurologically asymptomatic from brain metastases and has not received systemic corticosteroid therapy in the 10 days prior to beginning study intervention
* If capable of producing sperm, male participants agree to the following during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention. The length of time required to continue contraception for each study intervention is:
* Lenvatinib: 7 days
* Abstains from penile-vaginal intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agrees to remain abstinent. OR
* Uses contraception unless confirmed to be azoospermic
* Female participants are not pregnant or breastfeeding and are either not a woman of child-bearing potential (WOCBP) OR use a contraceptive method that is highly effective or are abstinent from heterosexual intercourse during the intervention period and for at least 120 days after the last dose of pembrolizumab or pembrolizumab/quavonlimab, or 30 days after the last dose of lenvatinib, whichever occurs last
* Has adequate organ function
* Female participants agree to abstain from breastfeeding during the study intervention period and for at least the time needed to eliminate study intervention after the last dose of study intervention. The length of time required for each study intervention is:
* MK-1308A: 120 days
* MK-3475: 120 days
* Lenvatinib: 30 days

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving immunosuppressive therapy within 10 days before the first dose of study intervention
* Has current or history of known leptomeningeal involvement
* Has received stereotactic or highly conformal radiotherapy within 2 weeks before the start of dosing
* Has clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study drug
* Has untreated or unresolved intracranial hemorrhage from central nervous system (CNS) metastasis
* Has an active infection requiring systemic therapy
* Has a known additional malignancy that is progressing or requires active treatment within the past 2 years
* Has ocular melanoma
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has known history of immunodeficiency virus (HIV)
* Has known history of hepatitis B or known hepatitis C virus
* Has a history of (noninfectious) pneumonitis that required steroids or current pneumonitis
* Has received prior systemic anticancer therapy within 4 weeks prior to randomization/allocation
* Has a history of whole brain irradiation
* Has received prior radiotherapy within 2 weeks of first dose of study intervention
* Has had major surgery <3 weeks prior to first dose of study intervention
* Has received a live or live attenuated vaccine within 30 days prior to the first dose of study intervention
* Has had an allogeneic tissue/solid organ transplant

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who experience an adverse event (AE) | Up to ~28 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience an AE will be reported.
Percentage of participants who discontinue study treatment due to an AE | Up to ~24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinue study treatment due to an AE will be reported.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) | Up to ~30 months
  ORR is defined as the percentage of participants in the analysis population who have a complete response (CR: disappearance of all target lesions) or partial response (PR: at ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters). Responses are according to RECIST 1.1 as assessed by blinded independent central review (BICR). RECIST 1.1 has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ.

SECONDARY OUTCOMES:
Duration of Response (DOR) per RECIST 1.1 | Up to ~30 months
  For participants in the analysis population who demonstrate a confirmed CR (disappearance of all target lesions) or confirmed PR (≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters), DOR is defined as the time from first documented CR or PR until progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of ≥1 new lesion is also considered PD. Responses are according to RECIST 1.1 as assessed by BICR. RECIST 1.1 has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Brain metastasis response rate (BMRR) per Response Assessment in Neuro- Oncology Brain Metastases (RANO-BM) | Up to ~30 months
  BMRR is defined as the percentage of participants in the analysis population who achieve a confirmed intracranial CR (disappearance of all lesions, no usage of corticosteroids and stable or improved clinical status) or PR (≥30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters, no progression of non-target lesions or new lesions, stable or decreased corticosteroid use, or stable or improved clinical status). Responses are according to RANO-BM as assessed by BICR. RANO-BM uses a combination of RECIST 1.1 and clinical data to assess response to treatment in brain metastases.
Brain metastasis duration of response (BM-DOR) per RANO-BM | Up to ~30 months
  For participants in the analysis population who demonstrate a confirmed intracranial CR (disappearance of all lesions, no usage of corticosteroids, stable or improved clinical status) or PR (≥30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters, no progression of non-target lesions or new lesions, stable or decreased corticosteroid use, or stable or improved clinical status), DOR is defined as the time from first documented CR or PR until PD or death due to any cause, whichever occurs first. Per RANO-BM, PD is defined as ≥20% increase in the sum of diameters of target lesions and an absolute increase of ≥5 mm in ≥1 lesion. Unequivocal increase in non-target lesions, the appearance of ≥1 new lesion or worsening of clinical status is also considered PD. Responses are according to RANO-BM as assessed by BICR. RANO-BM uses a combination of RECIST 1.1 and clinical data to assess response to treatment in brain metastases.
Progression-free survival (PFS) per RECIST 1.1 | Up to ~30 months
  PFS is defined as the time from randomization to the first documented PD or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Responses are according to RECIST 1.1 as assessed by BICR. RECIST 1.1 has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (36):
- United States (9):
  - The Angeles Clinic and Research Institute ( Site 4009), Los Angeles, California
  - UCLA Hematology & Oncology ( Site 4004), Los Angeles, California
  - Providence Saint John's Health Center ( Site 4010), Santa Monica, California
  - University of Colorado, Anschutz Cancer Pavilion ( Site 4012), Aurora, Colorado
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins ( Site 4022), Baltimore, Maryland
  - NYU Clinical Cancer Center ( Site 4002), New York, New York
  - Duke Cancer Institute ( Site 4005), Durham, North Carolina
  - Martha Morehouse Tower ( Site 4020), Columbus, Ohio
  - Inova Schar Cancer Institute ( Site 4011), Fairfax, Virginia
- Australia (2):
  - Calvary Mater Newcastle ( Site 4404), Waratah, New South Wales
  - Melanoma Institute Australia ( Site 4402), Wollstonecraft, New South Wales
- France (6):
  - Hopital La Timone ( Site 4103), Marseille, Bouches-du-Rhone
  - CHU de Bordeaux- Hopital Saint Andre ( Site 4108), Bordeaux, Gironde
  - Institut Claudius Regaud ( Site 4105), Toulouse, Haute-Garonne
  - Centre Hospitalier Lyon Sud ( Site 4102), Pierre-Bénite, Rhone
  - A.P.H. Paris, Hopital Saint Louis ( Site 4107), Paris
  - Gustave Roussy ( Site 4101), Villejuif, Île-de-France Region
- Israel (5):
  - HaEmek Medical Center ( Site 4703), Afula
  - Rambam Health Care Campus-Oncology ( Site 4704), Haifa
  - Hadassah Ein Karem Jerusalem ( Site 4702), Jerusalem
  - Rabin Medical Center-Oncology ( Site 4705), Petah Tikva
  - Chaim Sheba Medical Center ( Site 4701), Ramat Gan
- Italy (5):
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 4399), Milan
  - Istituto Europeo di Oncologia ( Site 4301), Milan
  - Istituto Nazionale Tumori Fondazione Pascale ( Site 4302), Napoli
  - Istituto Oncologico Veneto IRCCS ( Site 4355), Padua
  - Policlinico Le Scotte - A.O. Senese ( Site 4377), Siena
- South Africa (4):
  - CANCERCARE LANGENHOVEN DRIVE ONCOLOGY CENTRE ( Site 4865), Port Elizabeth, Eastern Cape
  - LIFE GROENKLOOF-Mary Potter Cancer Centre ( Site 4861), Pretoria, Gauteng
  - Sandton Oncology Medical Group (Pty) Ltd-Research ( Site 4863), Sandton, Gauteng
  - Cape Town Oncology Trials ( Site 4864), Cape Town, Western Cape
- Spain (2):
  - HOSPITAL CLÍNIC DE BARCELONA-ICHMO- Clinic Institut of Haematological and Oncological diseases ( Site 4801), Barcelona, Catalonia
  - Hospital Universitario Ramón y Cajal ( Site 4802), Madrid, Madrid, Comunidad de
- Switzerland (3):
  - Hôpitaux Universitaires de Genève (HUG)-Oncology ( Site 4603), Geneva, Canton of Geneva
  - CHUV Centre Hospitalier Universitaire Vaudois ( Site 4602), Lausanne, Canton of Vaud
  - Universitaetsspital Zuerich ( Site 4601), Zurich

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26250&tenant=MT_MSD_9011